CLINICAL TRIAL: NCT04203303
Title: Implications of the Human Microbiota for Health and Disease
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Principal Investigator, Mayo Clinic
Other Study IDs: 19-001234
Record Dates: First submitted 2019-10-11; First posted 2019-12-18 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Human Microbiota
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Observational
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The purpose of this study is to advance the understanding of human health and disease as it relates to environmental factors that may affect intestinal and non-intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Able to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients who are on the Mayo Clinic campus for clinic appointments or research study visits
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2030-10-15 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome Differences | 10 years
  compare the relative abundance of specific microorganism groups

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials